CLINICAL TRIAL: NCT06722066
Title: Impact of Aortic Annulus Calcification on Long-Term Outcomes Following Transcatheter Aortic Valve Replacement: Scientific Association of Interventional Cardiology - Transcatheter Aortic Valve Replacement (SAINT-TAVR) Calcium Registry
Brief Title: Impact of Aortic Annulus Calcification on Long-Term Outcomes Following Transcatheter Aortic Valve Replacement: SAINT-TAVR Calcium Registry
Acronym: SAINT-TAVR Ca
Status: Recruiting | Type: Observational
Sponsor: Eunpyeong St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Osung Kwon, Assistant professor, Eunpyeong St. Mary's Hospital
Other Study IDs: PC24OISI0131
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Transcatheter aortic valve replacement with ballon-expandable or self-expandable valves — Device: Edwards SAPIEN 3 valve, Medtronic Evolut valve, Boston Acurate Neo valve, or Abbott Navitor Access route: transfemorak, subclavian, transapical, transcarotid, or transcaval The use of balloon dilation will be left to the discretion of the operator.

SUMMARY:
The goal of this observational study is to learn about the long-term effects of aortic valve annular calcification in patients undergoing transcatheter aortic valve replacement (TAVR). The main question it aims to answer is:

Does the degree of aortic valve annular calcification prior to TAVR influence long-term clinical outcomes, including major adverse cardiovascular events including all-cause mortality, over a 3-year period?

Participants who have undergone TAVR as part of their regular medical care for severe aortic stenosis will have their pre-procedural imaging and clinical outcomes evaluated for a 3-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years or older.
2. Patients who have undergone transcatheter aortic valve replacement (TAVR) for severe aortic stenosis.
3. Individuals who have voluntarily provided written informed consent to participate.

Exclusion Criteria:

1. Individuals who have not provided written informed consent for this study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 19 years or older who have undergone transcatheter aortic valve replacement (TAVR) for severe aortic stenosis and have voluntarily expressed their willingness to participate through written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2031-12-02 (Estimated); Study Completion 2034-10-02 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 3 years follow-up

SECONDARY OUTCOMES:
Hospitalization for heart failure | 3 years follow-up
Stroke | 3 years follow-up
Myocardial infarction | 3 years follow-up
Permanent pacemaker insertion | 3 years follow-up
Vascular complication | 30 days follow-up

OTHER OUTCOMES:
Echo parameters | annual follow-up until 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Eunpyeong St. Mary's Hospital, College of Medicine, The Catholic University of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes